CLINICAL TRIAL: NCT07167979
Title: Investigating the Role of Neck Sensorimotor Integration and Eye Movement Training on Postural Control and Fall Risk in the Elderly
Brief Title: Neck Integration and Eye Movement Training for Fall Risk in the Elderly
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, PEI-CHI LIN, Principal Investigator, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20240131
Record Dates: First submitted 2025-08-20; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Elderly; Proprioception, Postural Balance; Oculomotor System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Strengthening Only (Placebo Comparator): The control group will receive an intervention consisting of neck muscle strengthening only.
  Interventions: Behavioral: Neck Strengthening Only
- Neck Strengthening plus Oculomotor Training (Experimental): The experimental group will receive an intervention combining neck muscle strengthening with oculomotor saccade tasks.
  Interventions: Behavioral: Combining neck muscle strengthening with oculomotor saccade tasks.

INTERVENTIONS:
Behavioral: Combining neck muscle strengthening with oculomotor saccade tasks. — he exercise program begins at 30% of 1RM, progressing by first increasing repetitions (8-10 up to 8-12) and then intensity (+5% of 1RM). Training sessions include a 5-minute warm-up, 20 minutes of exercise, and a 5-minute cool-down, performed twice per week for 30 minutes per session.
  Neck strengthening is performed using the Iron Neck, which provides constant resistance. Exercises include maintaining a neutral neck position, protraction-retraction, left-right rotation, dynamic figure-8 movements, and synchronized 360° head-body rotations. Each exercise consists of two sets of 8-12 repetitions, with 30 seconds rest between repetitions and 1 minute between sets.
  After neck training, participants in the intervention group perform oculomotor saccade tasks while maintaining a neutral head position. Five visual targets appear randomly in front of the participant for 1 second each. The task lasts 40 seconds, followed by 1-2 minutes of rest, and is repeated three times.
  Arms: Neck Strengthening plus Oculomotor Training
Behavioral: Neck Strengthening Only — he exercise program begins at 30% of 1RM, progressing by first increasing repetitions (8-10 up to 8-12) and then intensity (+5% of 1RM). Training sessions include a 5-minute warm-up, 20 minutes of exercise, and a 5-minute cool-down, performed twice per week for 30 minutes per session. Neck strengthening is performed using the Iron Neck, which provides constant resistance. Exercises include maintaining a neutral neck position, protraction-retraction, left-right rotation, dynamic figure-8 movements, and synchronized 360° head-body rotations. Each exercise consists of two sets of 8-12 repetitions, with 30 seconds rest between repetitions and 1 minute between sets.
  Arms: Neck Strengthening Only

SUMMARY:
Age is one of the primary risk factors for falls, with risk increasing as people get older. Research on fall risk and prevention has identified hundreds of contributing factors, showing that falls have complex and multifactorial causes. Risk factors can be categorized as environmental, extrinsic, or intrinsic. Intrinsic factors include physiological aspects-such as reduced lower-limb strength, impaired gait and balance, weaker grip strength, diminished sensory function, and poorer sensorimotor control-as well as psychological aspects, including fear of falling, depression, and cognitive decline. Strongly associated intrinsic risk factors include a history of falls, physical weakness, gait and balance disorders, certain medications, and dizziness. While fixed factors like age and fall history cannot be changed, identifying and targeting modifiable risk factors is crucial for prevention. Among these, gait and balance impairments are considered the most important modifiable intrinsic factors.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 to 85 years. Able to independently perform mobility necessary for activities of daily living.

No major medical conditions that significantly affect functional capacity.

Exclusion Criteria:

* Presence of central nervous system disorders (e.g., stroke). Severe musculoskeletal or visual injury of the lower limbs within the past three months that prevents participation in assessments.

Cognitive impairment. Current use of antidepressant medications.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Neck range of motion | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
Neck proprioception | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  Laser Joint Position Error Test
Neck position | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  Measurement Method: Craniovertebral Angle
Neck muscle | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  craniocervical flexion test, CCFT
Center of Pressure | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  force plate
Oculomotor | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  tobii eye tracker 5
  :Latency and Accuracy
Dynamic balance | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  y-balance
L/E Muscle strength | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  MicroFET2 MMT
Ankle proprioception | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  Joint Position Reproduction Test Kinesthesia
The Falls Efficacy Scale International | Assessments will be conducted at baseline, and at three, six, and twelve months post-intervention.
  The scale scores range from 16 to 64, with higher scores indicating greater severity

CONTACTS AND LOCATIONS:
Locations (1):
- Oculomotor training device, Kaohsiung City, Sanmin District, Taiwan